CLINICAL TRIAL: NCT01216800
Title: A Multicenter Randomized Study of Cochlear Sparing Intensity Modulated Radiotherapy Versus Conventional Radiotherapy in Patients With Parotid Tumors
Brief Title: Intensity-Modulated Radiation Therapy or 3-Dimensional Conformal Radiation Therapy in Decreasing Hearing Loss in Patients Who Have Undergone Surgery for Parotid Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000686212; ICR-CTSU/2007/10012; ISRCTN-81772291; EU-21073; MREC-05/Q0801/183; CRUK-08/004; ICR-RMH-2708
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Head and Neck Cancer; Ototoxicity; Radiation Toxicity
Keywords: ototoxicity; radiation toxicity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Ototoxicity; Radiation Injuries; Salivary Gland Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: assessment of therapy complications
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy is more effective in decreasing hearing loss in patients undergoing radiation therapy for parotid gland cancer.

PURPOSE: This randomized phase III trial is studying intensity-modulated radiation therapy to see how well it works compared with 3-dimensional conformal radiation therapy in decreasing hearing loss in patients who have undergone surgery for parotid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the potential of cochlear-sparing intensity-modulated radiotherapy (IMRT) versus conventional radiotherapy comprising 3-dimensional conformal radiotherapy in reducing the incidence of sensory-neural hearing loss in patients with parotid tumors undergoing radiotherapy to the parotid region.

Secondary

* To describe and compare the impact of both IMRT and conventional radiotherapy on physical, social and emotional well-being including generic functional and symptom aspects as well as disease-specific issues relevant to audiometry.

OUTLINE: This is a multicenter study. Patients are stratified according to center and radiotherapy dose. Patients are randomized to 1 of 2 treatment arms after surgical resection.

* Arm I (cochlear-sparing intensity-modulated radiotherapy [IMRT]): Patients undergo cochlear-sparing IMRT using the local planning system once daily, 5 days per week, for 6 weeks (total of 30 fractions) at a total dose of 60 Gy (65 Gy if macroscopic residual disease). Patients may undergo elective neck irradiation of the uninvolved lymph node areas once daily, 5 days per week, for 6 weeks.
* Arm II (conventional radiotherapy): Patients undergo conventional radiotherapy comprising 3-dimensional conformal radiotherapy once daily, 5 days per week, for 6 weeks (total of 30 fractions) at a total dose of 60 Gy (65 Gy if macroscopic residual disease). Patients may undergo elective neck irradiation of the uninvolved lymph node areas once daily, 5 days a week, for 5 weeks.

Patients complete quality-of-life questionnaires (EORTC QLQC30 v.3.0, the head and neck module H&N35, and a modified version of the Glasgow Hearing Aid Benefit profile) at baseline and at 6,12, 24, 36, 48, and 60 months after completion of study therapy. Patients also undergo audiological and vestibular assessment at 6 and 12 months following radiotherapy and then annually thereafter for up to 5 years.

After completion of study treatment, patients are followed up at 3, 6, 12, 18, and 24 months and then annually thereafter for up to 5 years (annually for recurrence for at least 10 years).

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant tumors of the parotid glands
* Adjuvant radiotherapy planned post-surgery
* No parotid tumors requiring primary radiotherapy
* No benign tumors requiring postoperative radiotherapy
* No metastases from squamous cell carcinoma of the head and neck to the parotid gland
* At high-risk of radiation-induced sensory-neural hearing loss with conventional radiotherapy due to the irradiation of the parotid bed to a dose equivalent of 60 Gy in 2 Gy/fraction with photon beams, using the wedge-pair technique

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* No hearing loss > 60 dB
* No previous or concurrent illness that, in the investigator's opinion, would interfere with either completion of therapy or follow-up
* Suitable to attend regular follow-up and undergo audiograms and toxicity monitoring and be available for long term follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the head and neck region
* No concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing sensory-neural hearing loss of at least 10 dB at bone conduction as assessed by audiograms at 4000 Hz one year after treatment

SECONDARY OUTCOMES:
Auditory assessment at 6 and 12 months following radiotherapy (RT) and then annually thereafter for up to 5 years
Vestibular assessment at baseline, at 6 and 12 months following RT, and then annually thereafter for up to 5 years
Quality of life at 6 and 12 months following RT and then annually thereafter for 5 years
Local and regional tumor control
Time to tumor progression
Overall survival
Acute and late side effects of RT as assessed by NCI CTCAE v 3.0 and the LENT SOMA and late RT scoring systems

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nutting, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom